CLINICAL TRIAL: NCT03490045
Title: Examining the Impact of an Intervention to Reduce Diaper Need and Increase Use of Pediatric Preventive Care
Brief Title: Intervention to Reduce Diaper Need and Increase Use of Pediatric Preventive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Diaper Bank Network (Unknown); Yale New Haven Health Primary Care Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000023616
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Diaper Dermatitis; Urinary Tract Infections; Infection; Depressive Symptoms; Stress
Keywords: Diaper Need; Well-Child Care; Infant Immunizations; Incentives; Basic Needs
MeSH Terms: conditions — Diaper Rash; Urinary Tract Infections; Infections; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): Postpartum women and their infants will be randomly assigned to the treatment condition and receive a diaper incentive for their participation.
  Interventions: Other: Diaper Incentive
- Comparison Condition (Active Comparator): Postpartum women and their infants will be randomly assigned to the control condition and will receive a conditional cash transfer of equivalent value of the diapers provided to the intervention group.
  Interventions: Other: Conditional Cash Transfer Condition

INTERVENTIONS:
Other: Diaper Incentive — A diaper incentive will be distributed to participants in the Intervention condition at 4-time points, which will coincide with the well-child visits that occur at 2-weeks, 2-months, 4-months, and 6-months. A follow-up assessment will also occur approximately 3 months after the family received their final distribution of diapers.
  Arms: Intervention Condition
Other: Conditional Cash Transfer Condition — Participants in the control condition will receive the cash equivalent value of the diapers distributed to the Experimental Condition for their participation at 4-time points, which will coincide with the well-child visits that occur at 2-weeks, 2-months, 4-months, and 6-months. A follow-up assessment will also occur approximately 3 months after the family received their final conditional cash transfer.
  Arms: Comparison Condition

SUMMARY:
Well-child care is the primary source of preventative health care for children. These visits provide an opportunity for physicians to assess an infant's biomedical health, development, and behavior, as well as help ensure timely immunizations, reduce the use of acute care services, and assess and family functioning. Yet, disparities in the utilization of pediatric care exist by race, ethnicity and income in the U.S., even despite high rates of overall access to primary care. Incentives have been proposed as one way to increase utilization of preventative care for mothers and children.

Diapering is another important form of preventative health care that can be particularly difficult for low-income parents due the cost of diapers, which is $70-80 per child per month, or approximately $960 per year, on average. And government programs, such as Special Supplemental Nutrition Program for Women, Infants, and Children (WIC), Supplemental Nutrition Assistance Program (SNAP), and Temporary Assistance for Needy Families (TANF), either cannot be used to purchase diapers, or do not provide enough assistance to cover the cost of diapers and other basic needs. A family's inability to provide an adequate supply of diapers for their child is called diaper need. Nationwide, one in three families with young children report experiencing diaper need, which was found to be significantly associated with maternal stress and depression, which in turn, can have a detrimental impact on a family's health and economic success.

The primary goal of this study is to conduct a randomized controlled trial of a diaper provision intervention designed to increase utilization of, and adherence to, well-child visits and reduce diaper need among low-resourced families in New Haven, CT.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial of a diaper incentive intervention whereby diapers will be used to achieve two separate but related aims.

First, diapers will be used as an incentive to increase utilization of, and adherence to, well-child visits, during the first year of a newborn's life. More specifically, postpartum women who receive care in the Yale New Haven Health System will be randomly assigned to receive a diaper incentive in conjunction with their attendance at regularly scheduled well-child visits, according to the American Academy of Pediatrics (AAP) recommended schedule during the first year of a child's life. Diapers will be provided at the completion of the 2- week, 2-month, 4- month and 6-month visits. A follow-up phone call assessment will also occur approximately 3 months after the family receives their final distribution of diapers or conditional cash transfer. Postpartum women randomly assigned to the control condition will receive the cash equivalent value of the diaper incentive for their participation at these same time points.

Second, diapers will be used to reduce the level of diaper need. This will be evaluated using a self-report diaper need survey that will be administered along with other surveys to women in the intervention and control conditions in accordance with the AAP well-child visit schedule. In addition to diaper need, the following domains will be assessed:

Depressive symptoms, perceived stress, maternal-child attachment, ability to meet basic needs, and demographic information including but not limited to race-ethnicity, mother's age, parity, marital status, education level, income, employment status, child(ren)'s sex, child(ren)'s age, health status, healthcare access, and use.

The investigators anticipate that this study will result in greater use of, and adherence to, the recommended schedule of pediatric well-child visits, as well as a greater reduction of diaper need among families in the intervention group. The investigators also anticipate that the reduction of diaper need will be associated with decreased parenting stress and improved diaper-related health among women and children, respectively, in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women who receive care at Yale New Haven Health
* Are about to give birth or recently gave birth to a singleton infant who is 0 to 1-week old (index child)
* Have not received a distribution of diapers for the index child
* English- speaking

Exclusion Criteria:

* Infant admitted to the NICU during the baseline assessment time period
* Infant admitted to the hospital at assessment visits 1-4
* Infant is born with or develops a gastrointestinal condition or illness that will impact the health outcomes of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Well-Child Visits | 9 Months
  The proportion of well-child visits attended.
Diaper Need | 9 Months
  The proportion of families that report experiencing diaper need. Diaper need will be measured via self-report using a scale developed by Smith et al.(2013).
Incidence of Diaper Dermatitis/Rash | 9 Months
  The number of episodes of diaper dermatitis/rash recorded by Yale New Haven Health physicians.
Incidence of Urinary Tract Infections | 9 Months
  The number of episodes of urinary tract infections (UTIs) recorded by Yale New Haven Health physicians.

SECONDARY OUTCOMES:
Depressive Symptoms Among Mothers | 9 Months
  A change in depressive symptom score between baseline and each time point. Depressive symptoms will be assessed using the Center for Epidemiologic Studies Depression Scale (CES-D)
Diaper-related Absences Among Mothers | 9 Months
  The proportion of mothers who report a decrease in diaper-related absences from work or school.
Stress | 9 Months
  A change in general stress scores between baseline and each time point. Stress will be measured by the Perceived Stress Scale 4 (PSS-4)
Basic Need | 9 Months
  Difference in basic need as measured by the U.S. Department of Agriculture Household Food Security Scale (2-item version) and Investigator-developed questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Wellbeing of Women and Mothers, 40 Temple Street, Ste 6B, Yale University, New Haven, Connecticut
  - Yale School of Medicine, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith MV, Kruse A, Weir A, Goldblum J. Diaper need and its impact on child health. Pediatrics. 2013 Aug;132(2):253-9. doi: 10.1542/peds.2013-0597. Epub 2013 Jul 29. PMID 23897910
- See also: Mental Health Outreach for MotherS Partnership — http://psychiatry.yale.edu/moms/haven/new.aspx